CLINICAL TRIAL: NCT06375746
Title: The Impact of a Customized Informative Video Prior to Induction of Labor on Anxiety Relieve - a Randomized Controlled Trial
Brief Title: The Impact of a Customized Informative Video Prior to Induction of Labor on Anxiety Relieve.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0091-22-WOMC
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Induction of Labor Affected Fetus / Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized video group (Experimental): In the video group patients will watch a personalized video prior to initiation of IOL in addition to standard counseling.
  Interventions: Other: Personalized video
- Control group (No Intervention): Patients will receive only standard counselling prior to initiation of IOL.

INTERVENTIONS:
Other: Personalized video — After enrollment and assignment to the intervention group, patients will receive a link to a personalized video describing the different induction methods by a text message.
  Other Names: Video group
  Arms: Personalized video group

SUMMARY:
To determine whether watching a personalized video prior to medically indicated labor induction among term parturients reduces anxiety levels according to the STAI questionnaire, compared to a standard counselling.

DETAILED DESCRIPTION:
The prevalence of induction of labor (IOL) has increased over the last decade, reaching between 15 to 30% of all deliveries in developed countries. IOL is commonly carried out using an extra-amniotic balloon (mechanical induction) or prostaglandins (pharmacological induction). Medical indications for IOL include maternal and fetal indications, where inducing labor results in improved maternal and neonatal outcomes compared with conservative management.

The process of labor induction can be associated with anxiety, especially in women undergoing IOL for the first time. Previous studies have focused on IOL success, examining the vaginal delivery rate or the time to delivery. Only a few studies have addressed the discomfort and anxiety that might accompany the procedures of IOL. A previous study from Australia found that women undergoing IOL wished to be presented with choice options, and receive more information about the process and its possible risks. A Swedish study found that the birth experience of women who underwent labor induction was less positive than that of women who gave birth spontaneously, with the former expressing greater concern for the baby's health.

Personalized video technology allows for the creation of a customized instructional videos, that may help reduce anxiety and decrease the element of uncertainty regarding IOL process and the expected fetal health. A possible advantage of this technology is that it may better engage patients and explain the medial intervention in a simple and clear manner. Many studies have examined the effect of presenting video clips, whether standardized or personalized, before medical procedures. These studies have shown significant effectiveness in improving adherence and strengthening the individual's commitment to the procedure, as well as creating a deeper understanding of the future events when using this technology. This technology is a simple method that does not involve pharmacological or invasive medical interventions to alleviate pain and anxiety.

The aim of this study is to examine whether using a personalized video reduces patients level of anxiety during induction of labor.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, aged 18-45, undergoing medical IOL at term.
* Unfavorable cervix (BISHOP score <6).
* Cervical ripening with either prostaglandin E2 (PGE2) tablets or extra-amniotic balloon (EAB).
* Provided consent to participate in the study.
* No language barrier preventing completion of the questionnaire.

Exclusion Criteria:

* Sensitivity to PGE2.
* Preterm labor.
* Premature rupture of membranes.
* Stillbirth.
* Elective pregnancy termination.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
STAI questionnaire score | Patient in both the study and the control groups will be asked to complete the STAI questionnaire twice as detailed below: • Prior to labor induction • After completion of IOL (either immediately after insertion of EAB or first PGE2 tablet).
  This is a validated questionnaire for the assessment of state anxiety called the State-Trait Anxiety Inventory (STAI). It includes 20 items presenting feelings characteristic of anxiety. Participants will be asked to rate how much each of the described feelings characterizes them at the moment on a scale ranging from 1 (not at all) to 4 (very much so). The final score on each questionnaire is obtained by summing all the ratings, after reversing the scale on the positively worded items. A higher score indicates a higher level of anxiety.

SECONDARY OUTCOMES:
satisfaction questionnaire | After completion of IOL (either immediately after insertion of EAB or first PGE2 tablet).
  Participants in both groups will be asked to complete a satisfaction questionnaire after IOL on a scale of one to five (1 - very low satisfaction, 2 - low satisfaction, 3 - moderate satisfaction, 4 - high satisfaction, 5 - very high satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goffinet F, Dreyfus M, Carbonne B, Magnin G, Cabrol D. [Survey of the practice of cervical ripening and labor induction in France]. J Gynecol Obstet Biol Reprod (Paris). 2003 Nov;32(7):638-46. French. PMID 14699333
- [Background] Mackenzie IZ. Induction of labour at the start of the new millennium. Reproduction. 2006 Jun;131(6):989-98. doi: 10.1530/rep.1.00709. PMID 16735538
- [Background] Declercq ER, Sakala C, Corry MP, Applebaum S. Listening to Mothers II: Report of the Second National U.S. Survey of Women's Childbearing Experiences: Conducted January-February 2006 for Childbirth Connection by Harris Interactive(R) in partnership with Lamaze International. J Perinat Educ. 2007 Fall;16(4):15-7. doi: 10.1624/105812407X244778. PMID 18769522
- [Background] National Collaborating Centre for Women and Children'sHealth. Induction of labour. London: NICE, 2008
- [Background] Public Health Agency of Canada. Canadian Perinatal Health Report, 2008 edn. Ottawa: Public Health Agency of Canada, 2008
- [Background] Mozurkewich EL, Chilimigras JL, Berman DR, Perni UC, Romero VC, King VJ, Keeton KL. Methods of induction of labour: a systematic review. BMC Pregnancy Childbirth. 2011 Oct 27;11:84. doi: 10.1186/1471-2393-11-84. PMID 22032440
- [Background] Nuutila M, Halmesmaki E, Hiilesmaa V, Ylikorkala O. Women's anticipations of and experiences with induction of labor. Acta Obstet Gynecol Scand. 1999 Sep;78(8):704-9. PMID 10468063
- [Background] Kleiner I, Mor L, Friedman M, Abeid AA, Shoshan NB, Toledano E, Bar J, Weiner E, Barda G. The use of virtual reality during extra-amniotic balloon insertion for pain and anxiety relief-a randomized controlled trial. Am J Obstet Gynecol MFM. 2024 Jan;6(1):101222. doi: 10.1016/j.ajogmf.2023.101222. Epub 2023 Nov 10. PMID 37951577